CLINICAL TRIAL: NCT03809949
Title: Opioid Free Versus Opioid Balanced Anesthesia in Middle Ear Surgery.
Brief Title: Opioid Free Versus Opioid Balanced Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050108073(18/12/2018)
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: PONV; Opioid Use
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: To compare between opioid and opioid free anaesthesia on post-operative nausea and vomiting in middle ear surgery
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Doctors, patients and outcomes assessors will be blinded regarding the technique used in anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl Opioid Anesthesia (Active Comparator): Fentanyl (1mg/kg i.v.) will be administered before general anaesthesia (GA). GA will be maintained with inhalation anaesthetics (isoflurane) at a minimum alveolar concentration of 0.7-1.3.
  Interventions: Drug: Fentanyl Opioid anesthesia
- Saline Nonopioid Anesthesia (Placebo Comparator): Opioid free anesthesia (syringe of saline is given instead of fentanyl) and the same general anesthesia is given as group A(muscle relaxant ,propofol, inhalation for maintance).
  Interventions: Drug: Saline Nonopioid anesthesia

INTERVENTIONS:
Drug: Fentanyl Opioid anesthesia — To compare between opioid and opioid free anaesthesia on post-operative nausea and vomiting in middle ear surgery
  Arms: Fentanyl Opioid Anesthesia
Drug: Saline Nonopioid anesthesia — To compare between opioid and opioid free anaesthesia on post-operative nausea and vomiting in middle ear surgery
  Arms: Saline Nonopioid Anesthesia

SUMMARY:
OPIOID FREE VERSUS OPIOID BALANCED ANAESTHESIA IN MIDDLE EAR SURGERY AIM OF THE WORK

Primary aim:

To compare between opioid and opioid free anaesthesia on post-operative nausea and vomiting in middle ear surgery

Secondary aim:

Monitoring analgesia, post-operative satisfaction and drowsiness.

DETAILED DESCRIPTION:
After approval of the Ethical Committee of Faculty of Medicine, Alexandria University and having an informed written consent from every patient included in the study, the present study will be carried out in Alexandria Main University Hospitals on sixty adult patients belonging to ASA class I or II scheduled for middle ear surgery under general anaesthesia.

(The sample size is approved to be sufficient by the Department of Statistics, Medical Research Institute, University of Alexandria).

Inclusion criteria:

* Patients of either sex.
* American Society Anesthesiologists' physical status I-II.
* Age between 18 and 50 years. Exclusion criteria:(depend on table 1)
* Patients with gastrointestinal disease.
* A history of motion sickness, or a previous episode of PONV.
* Patient received any opioid, steroid, or antiemetic medication within 72 h before surgery.
* Those who were pregnant or menstruating.
* History of opioid or drug abuse. METHODS Patients will be randomly allocated into two equal groups (thirty patients each) using the closed envelope method.

I will compare postoperative nausea and vomiting (PONV) in patients scheduled for middle ear surgery. Sixty patients will be randomly allocated to receive either balanced anaesthesia (group A) using fentanyl, propofol and isoflurane, or opioid free anaesthesia (group B) using propofol and isoflurane. Pain scores, nausea ⁄ vomiting scores, conditions for surgery and analgesic requirements will be recorded post operatively.

Anaesthetic management Preoperative management

All patients will be visited before surgery to be clinically assessed and the preoperative surveillance includes:

* Haematological screening (Complete blood picture, Serum electrolytes).
* Standard coagulation studies e.g. prothrombin time, international normalized ratio (PT-INR).

On arrival to the operating room and before anaesthetic induction all patients will be monitored by the standard routine monitoring, which include:

* A 5-lead electrocardiography.
* A non-invasive blood pressure (NIBP) (mmHg).
* Pulse oximetry (%).
* Capnography. (End Tidal CO2 pattern and value in mmHg).
* Temperature monitoring. A peripheral intravenous cannula of 20 gauges will be inserted in a dorsal vein of the non-dominant hand.

Premedication with Midazolam in a dose of 0.02mg/ Kg will be used. Induction Preoxygenation with 100 % O2 for 3 minutes. General anaesthesia will be induced by propofol (2 mg/kg) and atracurium (0.5 mg/kg) intravenously guided by a nerve stimulator, followed by endotracheal intubation after loss of train of four.

All the patients will receive i.v. acetaminophen (1000 mg) _20 min after induction and i.v. ketorolac (30 mg).

Local analgesia will be injected by surgeon. All patients will receive beta blocker (Inderal 1mg) and magnesium sulphate (15-30mg/kg) for achieving hypotensive anaesthesia.

Maintenance Maintenance of general anaesthesia with a mixture of isoflurane (1MAC) and oxygen.

All patients will be mechanically ventilated with an anaesthesia machine to keep SpO2 > 95% and end-tidal CO2 between 35-45 mmHg.

Additional atracurium will be administrated as appropriate in bolus doses if needed.

Group A Fentanyl (1mg/kg i.v.) will be administered before general anaesthesia (GA). GA will be maintained with inhalation anaesthetics (isoflurane) at a minimum alveolar concentration of 0.7-1.3.

Group B Opioid free anesthesia (syringe of saline is given instead of fentanyl) and the same general anesthesia is given as group A(muscle relaxant ,propofol, inhalation for maintance).

Recovery At the end of surgery, isoflurane will be discontinued, 100% oxygen will be given, all patients will be planned for extubation in the operating room depending on recovery criteria after complete reversal of muscle relaxant with neostigmine (up to 5 mg).

Tracheal extubation will be performed in a semi- sitting position after fulfilling the criteria for extubation. Extubation criteria include: a fully conscious patient, haemodynamic stability, reversal of neuromuscular blockade, TOF ratio 0.9 - 1 on nerve stimulator, and the ability of head lift for 5 seconds.

Postoperative multimodal pain management Postoperative pain will be treated with i.v. acetaminophen (1000mg) and i.v. ketorolac (30 mg) every 6 h for the first 24 h. Postoperative pain will be measured on an 11-point numeric pointscale (NPS).

management of PONV Dexamethasone (8 mg i.v.) will be administered during induction, ondansetron (4 mg i.v.) and metoclopramide (10 mg i.v.) post operative if Patients complaining of PONV after discharge from the PACU.

Measurements

1. Demographic data:

   Age (years), sex, weight (kilograms).
2. Hemodynamic parameters:

   * Pulse oximetry (%)
   * Heart rate (HR). Beats/minute
   * Mean Non-Invasive arterial blood pressure (NIBP) (mmHg)
3. Pain assessment The level of pain will be assessed on an 11-point NPS. Patients will be asked to determine their own 'acceptable' pain score.

   The 11-point numeric scale ranges from '0' representing no pain extreme to '10' representing the other pain extreme (worst pain imaginable).(8)
4. Nausea and vomiting assessment (table2,3) Patients will be asked to rate the worst episode of PONV on a four-point verbal rating scale (VRS) (none, mild, moderate, or severe). Patients were also will be asked whether they experienced retching or vomiting.
5. Sedation assessment

Sedation score:

0. Alert

1. Mild, drowsy, easy to awake
2. Moderate, easy to arouse
3. Severe: somnolent difficult to arouse
4. Sleeping The Sedation score will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours.

6. Satsifacation of patient assessment by QoR40 questionnaire The QoR-40 is a global measure of quality of recovery. It incorporates five dimensions: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).(29) Timing Hemodynamic (blood pressure, pulse) of Patients will be assessed during the surgery every 10 minutes and at 1 and 2 h after the end of surgery and at discharge from the day unit. At each of these times, the nurse recorded the incidence and worst severity of pain, nausea and emesis since the last evaluation using the same criteria as before. Any medication will be given for pain or nausea (administered for moderate-severe symptoms, or at patient request) will be also recorded, till the time of discharge. Patients will be discharged with medication comprising slow-release ibuprofen. The following day, the researcher will telephone the patient to assess the incidence and worst severity of pain, nausea and emesis since discharge and whether any analgesia or antiemetics will be taken. Patients will be also asked to record their satisfaction with the control of pain, the control of sickness and their overall day surgery experience on 11-point (0-10) verbal rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex.
* American Society Anesthesiologists' physical status I-II.
* Age between 18 and 50 years.

Exclusion Criteria:

* Patients with gastrointestinal disease.
* A history of motion sickness, or a previous episode of PONV.
* Patient received any opioid, steroid, or antiemetic medication within 72 h before surgery.
* Those who were pregnant or menstruating.
* History of opioid or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
PONV | 72 hours
  Post operative nausea and vomiting from 0-3 for nausea and 0 to 4 for vomiting

SECONDARY OUTCOMES:
analgesia.post-operative pain | 72 hours
  analgesia, post-operative VAS score
Patient satisfaction | 72 hours
  satisfaction degree by QoR40 questionnaire from 40 to 200
Drowsiness | 72 hours
  Drowsiness scores by RAMSY sedation score from 0 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quemby DJ. Day surgery development and practice: key factors for a successful pathway. CEACCP 2014;14: 256-61.
- [Background] Moore KL, Dalley AF. Clinically orientated anatomy. 4th ed. Philadelphia: Lippinocott Williams & Wilkins; 1999.
- [Background] Dhillon RS, East CA. Ear, nose, throat, and head and neck surgery: an illustrated colored text. 2nd ed. New York, Edinburgh: Churchill Livingstone;1999
- [Background] Deacock AR. Aspects of anaesthesia for middle ear surgery an blood loss during stapedectomy. Proc R Soc Med. 1971 Dec;64(12):1226-8. doi: 10.1177/003591577106401226. No abstract available. PMID 4399792
- [Background] Miller RD. Miller's anesthesia, 6th ed. Vol 2. New York: Elsevier/Churchill Livingstone; 2005.
- [Background] Morgan EG, Mikhail MS, Murray MJ. Clinical anesthesiology. 4th ed. New York: Lange Medical Books/McGraw-Hill; 2006.
- [Background] Bailey CR. Management of outpatient ear, nose and throat surgery. Curr Opin Anaesthesiol. 2001 Dec;14(6):617-21. doi: 10.1097/00001503-200112000-00003. PMID 17019154
- [Background] Honkavaara P, Saarnivaara L, Klemola UM. Prevention of nausea and vomiting with transdermal hyoscine in adults after middle ear surgery during general anaesthesia. Br J Anaesth. 1994 Dec;73(6):763-6. doi: 10.1093/bja/73.6.763. PMID 7880660
- [Background] Fujii Y, Toyooka H, Tanaka H. Prophylactic antiemetic therapy with a combination of granisetron and dexamethasone in patients undergoing middle ear surgery. Br J Anaesth. 1998 Nov;81(5):754-6. doi: 10.1093/bja/81.5.754. PMID 10193289 (Retraction: PMID 23508503 Br J Anaesth. 2013 Apr;110(4):669)
- [Background] Fujii Y, Saitoh Y, Tanaka H, Toyooka H. Anti-emetic efficacy of prophylactic granisetron compared with perphenazine for the prevention of post-operative vomiting in children. Eur J Anaesthesiol. 1999 May;16(5):304-7. doi: 10.1046/j.1365-2346.1999.00483.x. PMID 10390665 (Retraction: PMID 23571441 Eur J Anaesthesiol. 2013 May;30(5):263)
- [Background] Gombar S, Kaur J, Kumar Gombar K, Dass A, Singh A. Superior anti-emetic efficacy of granisetron-dexamethasone combination in children undergoing middle ear surgery. Acta Anaesthesiol Scand. 2007 May;51(5):621-4. doi: 10.1111/j.1399-6576.2007.01296.x. PMID 17430326
- [Background] Bovill JG, Sebel PS, Stanley TH. Opioid analgesics in anesthesia: with special reference to their use in cardiovascular anesthesia. Anesthesiology. 1984 Dec;61(6):731-55. PMID 6150663
- [Background] Long DR, Lihn AL, Friedrich S, Scheffenbichler FT, Safavi KC, Burns SM, Schneider JC, Grabitz SD, Houle TT, Eikermann M. Association between intraoperative opioid administration and 30-day readmission: a pre-specified analysis of registry data from a healthcare network in New England. Br J Anaesth. 2018 May;120(5):1090-1102. doi: 10.1016/j.bja.2017.12.044. Epub 2018 Mar 9. PMID 29661386
- [Background] Golembiewski J, Chernin E, Chopra T. Prevention and treatment of postoperative nausea and vomiting. Am J Health Syst Pharm. 2005 Jun 15;62(12):1247-60; quiz 1261-2. doi: 10.1093/ajhp/62.12.1247. PMID 15947124
- [Background] Macario A, Weinger M, Truong P, Lee M. Which clinical anesthesia outcomes are both common and important to avoid? The perspective of a panel of expert anesthesiologists. Anesth Analg. 1999 May;88(5):1085-91. doi: 10.1097/00000539-199905000-00023. PMID 10320175
- [Background] Smith I, Terhoeve PA, Hennart D, Feiss P, Harmer M, Pourriat JL, Johnson IA. A multicentre comparison of the costs of anaesthesia with sevoflurane or propofol. Br J Anaesth. 1999 Oct;83(4):564-70. doi: 10.1093/bja/83.4.564. PMID 10673870
- [Background] Smith I, Thwaites AJ. Target-controlled propofol vs. sevoflurane: a double-blind, randomised comparison in day-case anaesthesia. Anaesthesia. 1999 Aug;54(8):745-52. doi: 10.1046/j.1365-2044.1999.00953.x. PMID 10460526
- [Background] Fleischmann E, Akca O, Wallner T, Arkilic CF, Kurz A, Hickle RS, Zimpfer M, Sessler DI. Onset time, recovery duration, and drug cost with four different methods of inducing general anesthesia. Anesth Analg. 1999 Apr;88(4):930-5. doi: 10.1097/00000539-199904000-00046. PMID 10195551
- [Background] Fredman B, Nathanson MH, Smith I, Wang J, Klein K, White PF. Sevoflurane for outpatient anesthesia: a comparison with propofol. Anesth Analg. 1995 Oct;81(4):823-8. doi: 10.1097/00000539-199510000-00028. PMID 7574017
- [Background] Shakir AAK, Ramachandra V, Hasan MA. Day surgery postoperative nausea and vomiting at home related to preoperative fentanyl. J One-day Surg 1997;6:10-1.
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Vandermeulen EP. Controlling the stress response. In: White PF (ed). Textbook of Intravenous Anesthesia. Baltimore: Williams & Wilkins; 1997. p. 565-79.
- [Background] Borgeat A, Wilder-Smith OH, Saiah M, Rifat K. Subhypnotic doses of propofol possess direct antiemetic properties. Anesth Analg. 1992 Apr;74(4):539-41. doi: 10.1213/00000539-199204000-00013. PMID 1554120
- [Background] Gan TJ, Glass PSA. Balanced anesthesia. In: White PF (ed). Textbook of Intravenous Anesthesia. Baltimore: Williams & Wilkins; 1997. p. 347-74.
- [Background] Smith I. Inhalational anesthetic agents. In: Hemmings HC, Hopkins PM (eds). Foundations of Anesthesia. 2nd ed. London: Elsevier; 2005. p. 311-21.
- [Background] Ziemann-Gimmel P, Goldfarb AA, Koppman J, Marema RT. Opioid-free total intravenous anaesthesia reduces postoperative nausea and vomiting in bariatric surgery beyond triple prophylaxis. Br J Anaesth. 2014 May;112(5):906-11. doi: 10.1093/bja/aet551. Epub 2014 Feb 18. PMID 24554545
- [Background] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031
- [Background] Feld JM, Hoffman WE, Stechert MM, Hoffman IW, Ananda RC. Fentanyl or dexmedetomidine combined with desflurane for bariatric surgery. J Clin Anesth. 2006 Feb;18(1):24-8. doi: 10.1016/j.jclinane.2005.05.009. PMID 16517328
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753